CLINICAL TRIAL: NCT06118437
Title: Establishment and Validation of a Clinical Predictive Model for Gastrointestinal Cancer Screening Based on Patient-related Risk Factors: a Prospective, Multicenter Cross-sectional Study
Brief Title: Establishment and Validation of a Clinical Predictive Model for Gastrointestinal Cancer Screening Based on Patient-related Risk Factors
Status: Recruiting | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, professor, Air Force Military Medical University, China
Other Study IDs: XJLL-KY-20232231
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2024-07

CONDITIONS: Malignant Tumor of Digestive Tract; Risk Factors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gastrointestinal tumors (esophageal cancer, gastric cancer, colorectal cancer) seriously threaten human health, with a high incidence rate and cancer related hope mortality. Digestive endoscopy is the main method for screening gastrointestinal tumors. Early screening of gastrointestinal tumors can improve the detection of early cancer and improve prognosis. The five-year survival rate of early stage tumors after comprehensive treatment can reach 90%, while the five-year survival rate of late stage tumors is less than 30%. Therefore, the screening of gastrointestinal tumors is very important.

Studies have shown that there are similarities in risk factors for gastrointestinal tumors, such as age, gender, family history, smoking, alcohol consumption, etc. Currently, established digestive malignancies are targeted at a single malignant tumor. At present, there is a lack of understanding of the overall risk factors associated with gastrointestinal tumors and the establishment of relevant risk prediction models.

Therefore, we conducted a prospective, multicenter cross-sectional study to explore the independent risk factors of combined gastrointestinal tumors and establish a risk prediction model for combined screening of gastrointestinal tumors.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-80;
* Undergoing both gastroscopy and colonoscopy simultaneously.

Exclusion Criteria:

* History of esophageal, gastric, or colorectal cancer;
* Suspicions of gastrointestinal obstruction or perforation;
* History of gastrointestinal tract surgery;
* Not suitable for endoscopic examination due to serious diseases or unstable hemodynamics;
* Unavailable relevant information;
* Pregnancy or lactation period;
* Unavailable informed consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Continuous patients who underwent both gastroscopy and colonoscopy at the digestive endoscopy center from October 2023 to May 2025
Sampling Method: Non-Probability Sample
Enrollment: 1550 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Overall detection rate of gastrointestinal cancer | 2 years
  The proportion of at least one type of gastrointestinal malignant tumor detected

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing of Digestive Diseases, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Klein EA, Richards D, Cohn A, Tummala M, Lapham R, Cosgrove D, Chung G, Clement J, Gao J, Hunkapiller N, Jamshidi A, Kurtzman KN, Seiden MV, Swanton C, Liu MC. Clinical validation of a targeted methylation-based multi-cancer early detection test using an independent validation set. Ann Oncol. 2021 Sep;32(9):1167-1177. doi: 10.1016/j.annonc.2021.05.806. Epub 2021 Jun 24. PMID 34176681